CLINICAL TRIAL: NCT05515263
Title: Snack Foods and Their Impact on Immune Optimisation to the Influenza Vaccination: a Randomised Controlled Trial of a Vaccination Model of Immune Response
Brief Title: Snack Foods and Their Impact on the Immune Response Following Influenza Vaccination
Acronym: NutrImmune
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HR/DP-21/22-33040
Record Dates: First submitted 2022-08-17; First posted 2022-08-25 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Immune Response
Keywords: Immune Response; Immune Function; Gut Health; Gut Microbiota; Snack

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention snack (Experimental): The intervention group will receive a snack food believed to be beneficial for immune function (high content of immunoregulatory nutrients).
  Interventions: Dietary Supplement: Intervention snack
- Control snack (Placebo Comparator): The control group will receive an isocaloric, commercially available snack food (low content of immunoregulatory nutrients).
  Interventions: Dietary Supplement: Control snack

INTERVENTIONS:
Dietary Supplement: Intervention snack — To be eaten in replacement of usual snacks twice a day for 8 weeks.
  Arms: Intervention snack
Dietary Supplement: Control snack — To be eaten in replacement of usual snacks twice a day for 8 weeks.
  Arms: Control snack

SUMMARY:
The purpose of this study is to evaluate the impact of replacing usual snacks with alternative snack foods on the immune response to influenza vaccination in a population of healthy, middle-aged adults.

DETAILED DESCRIPTION:
Nutrition plays an important role in the immune system by providing energy and metabolites to support the function of immune cells, allowing them to initiate effective immune responses. Diet is therefore a modifiable factor in impacting immune function and is currently a topic of substantial interest in health research. Snack consumption has been shown to account for approximately 20-30% of daily energy intake in adults. Therefore, snack choices have the potential to influence dietary intake and quality, and therefore immune function, both positively and negatively. This study assesses the effect of replacing usual snacks with alternative snack foods on the immune response in a model of viral infection - the seasonal influenza vaccine containing four prevalent influenza virus strains for the 2022/23 or 2023/24 influenza season, as determined by the World Health Organization.

This study is a parallel group, randomised controlled trial that will examine the replacement of usual snack foods with alternative snack foods on the immune response to seasonal influenza vaccination in humans, which will be assessed by measuring rates of seroconversion, and other immunological markers following vaccination. The intervention will be for 8 weeks, and influenza vaccination will be administered at 4-week midpoint. Participants will be followed up 3 months post-vaccination to assess incidence of upper respiratory symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women, aged between 40-64 years
2. Body mass index (BMI) of 18.50 - 29.99 kg/m2
3. Individuals who regularly consume snacks (≥2 per day, excluding fruit, vegetable, nut and seed snacks)
4. Fibre intake <30 g/d
5. Willing to avoid receiving any vaccination (except for COVID-19 vaccination) from one month prior to the baseline visit until completion of the 8-week intervention period
6. Willing to avoid receiving any COVID-19 vaccination/booster between week 2 and week 8 of the intervention period
7. Willing to discontinue use of prebiotics and probiotics during the trial
8. Willing to follow the protocol and provide consent

Exclusion Criteria:

1. Allergy or intolerance to any intervention products
2. Dislike of any intervention products
3. Immunodeficiency/immunosuppression due to disease or medication, such as:

   * Chronic inflammatory disease or autoimmune disease (e.g., rheumatoid arthritis, inflammatory bowel disease, psoriasis) or primary or secondary immunodeficiency disease (e.g., HIV infection)
   * Ongoing therapy with immunomodulators or immunosuppressants (e.g., chemotherapy, oral corticosteroids, daily use of inhaled or nasal corticosteroids)
   * Other immunodeficient state (e.g., asplenia).
4. Medical history of any of the following: diabetes, major active psychiatric conditions (e.g. schizophrenia), current eating disorder, alcohol abuse, active treatment for cancer in the last year, severe neurological, endocrine, renal, cardiac or pulmonary disease (or any other chronic medical condition), severe oesophagitis, gastritis or duodenitis, active diverticulitis or intestinal/colonic strictures, Coeliac disease, Crohn's disease or Ulcerative colitis, stem cell or organ transplant, gut resection surgery, bleeding disorder, anaphylaxis or any other major or chronic condition known to impact study outcome measures.
5. Ongoing use of antiviral agents, or any other drugs known to impact study outcome measures
6. Use of immunoglobulins and/or any blood products within the three months prior to vaccination
7. Ongoing use of anticoagulants (e.g., warfarin)
8. Antibiotic treatment in the month prior to the start of the study
9. Consumption of probiotics or prebiotic products within the four weeks prior to the start of the study
10. History of severe adverse reaction and/or allergic reaction associated with the influenza vaccine or any other vaccine
11. Known allergy or hypersensitivity to any component of the vaccine including: sodium chloride, potassium chloride, magnesium chloride hexahydrate, disodium phosphate dihydrate, potassium dihydrogen phosphate; and possible trace residues: beta-propiolactone, cetyltrimethylammonium bromide, and polysorbate 80
12. Suffered from influenza illness in the six months prior to the start of the study
13. For participants recruited on or before 30/06/2023, exclusion criteria is: already vaccinated with any influenza vaccine licensed for the 2022/2023 season; For participants recruited after 30/06/2023, exclusion criteria is: already vaccinated with any influenza vaccine licensed for the 2023/2024 season
14. Received any influenza vaccination within six months prior to the start of the study
15. Received any other vaccinations within one month prior to the start of the study (except for COVID-19 vaccination)
16. Women who are pregnant, lactating or planning pregnancy
17. Ongoing alcohol, drug or medication abuse
18. Unexplained or unintentional weight loss in the past six months

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Rates of seroconversion for ≥1 influenza virus strain | Week 8
  The proportion of participants achieving seroconversion (≥4-fold increase in specific antibody titre) in at least one influenza virus strain. Titres will be assessed using the Hemagglutination Inhibition Assay (HAI) and fold change will be calculated.

SECONDARY OUTCOMES:
Rates of seroconversion for A/Wisconsin/588/2019 (H1N1)pdm09-like virus strain (strain 1a) | Week 8
  The proportion of participants achieving seroconversion for A/Wisconsin/588/2019 (H1N1)pdm09-like virus strain. Titres will be assessed by HAI and fold change will be calculated.
Rates of seroconversion for A/Wisconsin/67/2022 (H1N1)pdm09-like virus strain (strain 1b) | Week 8
  The proportion of participants achieving seroconversion for A A/Wisconsin/67/2022 (H1N1)pdm09-like virus strain. Titres will be assessed by HAI and fold change will be calculated.
Rates of seroconversion for A/Darwin/6/2021 (H3N2)-like virus strain (strain 2) | Week 8
  The proportion of participants achieving seroconversion for A/Darwin/6/2021 (H3N2)-like virus strain. Titres will be assessed by HAI and fold change will be calculated.
Rates of seroconversion for influenza virus B/Austria/1359417/2021 (B/Victoria lineage)-like virus strain (strain 3) | Week 8
  The proportion of participants achieving seroconversion for B/Austria/1359417/2021 (B/Victoria lineage)-like virus strain. Titres will be assessed by HAI and fold change will be calculated.
Rates of seroconversion for B/Phuket/3073/2013 (B/Yamagata lineage)-like virus strain (strain 4) | Week 8
  The proportion of participants achieving seroconversion for B/Phuket/3073/2013 (B/Yamagata lineage)-like virus strain. Titres will be assessed by HAI and fold change will be calculated.
Proportion of participants who do not achieve seroconversion for any influenza virus strain | Week 8
  Titres will be assessed by HAI and fold change will be calculated.
Rates of seroconversion for only 1 influenza virus strain | Week 8
  The proportion of participants achieving seroconversion for 1 influenza virus strain. Titres will be assessed by HAI and fold change will be calculated.
Rates of seroconversion for 2 influenza virus strains | Week 8
  The proportion of participants achieving seroconversion for 2 influenza virus strains. Titres will be assessed by HAI and fold change will be calculated.
Rates of seroconversion for 3 influenza virus strains | Week 8
  The proportion of participants achieving seroconversion for 3 influenza virus strains. Titres will be assessed by HAI and fold change will be calculated.
Rates of seroconversion for 4 influenza virus strains | Week 8
  The proportion of participants achieving seroconversion for all 4 influenza virus strains. Titres will be assessed by HAI and fold change will be calculated.
Geometric mean antigen-specific titres for or A/Wisconsin/588/2019 (H1N1)pdm09-like virus strain (strain 1a) | Week 0, 4 and 8
  Titres will be assessed by HAI.
Geometric mean antigen-specific titres for A/Wisconsin/67/2022 (H1N1)pdm09-like virus strain (strain 1b) | Week 0, 4 and 8
  Titres will be assessed by HAI.
Geometric mean antigen-specific titres for A/Darwin/6/2021 (H3N2)-like virus strain (strain 2) | Week 0, 4 and 8
  Titres will be assessed by HAI.
Geometric mean antigen-specific titres for B/Austria/1359417/2021 (B/Victoria lineage)-like virus strain (strain 3) | Week 0, 4 and 8
  Titres will be assessed by HAI.
Geometric mean antigen-specific titres for B/Phuket/3073/2013 (B/Yamagata lineage)-like virus strain (strain 4) | Week 0, 4 and 8
  Titres will be assessed by HAI assay.
Fold change in antigen-specific titres for A/Wisconsin/588/2019 (H1N1)pdm09-like virus strain (strain 1a) | Week 8
  Titres will be assessed by HAI and fold change will be calculated.
Fold change in antigen-specific titres for A/Wisconsin/67/2022 (H1N1)pdm09-like virus strain (strain 1b) | Week 8
  Titres will be assessed by HAI and fold change will be calculated.
Fold change in antigen-specific titres for A/Darwin/6/2021 (H3N2)-like virus strain (strain 2) | Week 8
  Titres will be assessed by HAI and fold change will be calculated.
Fold change in antigen-specific titres for B/Austria/1359417/2021 (B/Victoria lineage)-like virus strain (strain 3) | Week 8
  Titres will be assessed by HAI and fold change will be calculated.
Fold change in antigen-specific titres for B/Phuket/3073/2013 (B/Yamagata lineage)-like virus strain (strain 4) | Week 8
  Titres will be assessed by HAI and fold change will be calculated.
Seroprotection for ≥1 influenza virus strain | Week 8
  The proportion of participants achieving seroprotection (HAI titre of ≥1:40) in at least one of the four influenza virus strains.
Seroprotection for A/Wisconsin/588/2019 (H1N1)pdm09-like virus strain (strain 1a) | Week 8
  The proportion of participants achieving seroprotection (HAI titre of ≥1:40) for A/Wisconsin/588/2019 (H1N1)pdm09-like virus strain.
Seroprotection for A/Wisconsin/67/2022 (H1N1)pdm09-like virus strain (strain 1b) | Week 8
  The proportion of participants achieving seroprotection (HAI titre of ≥1:40) for A/Wisconsin/67/2022 (H1N1)pdm09-like virus strain.
Seroprotection for A/Darwin/6/2021 (H3N2)-like virus strain (strain 2) | Week 8
  The proportion of participants achieving seroprotection (HAI titre of ≥1:40) for A/Darwin/6/2021 (H3N2)-like virus strain.
Seroprotection for B/Austria/1359417/2021 (B/Victoria lineage)-like virus strain (strain 3) | Week 8
  The proportion of participants achieving seroprotection (HAI titre of ≥1:40) for B/Austria/1359417/2021 (B/Victoria lineage)-like virus strain.
Seroprotection for B/Phuket/3073/2013 (B/Yamagata lineage)-like virus strain (strain 4) | Week 8
  The proportion of participants achieving seroprotection (HAI titre of ≥1:40) for B/Phuket/3073/2013 (B/Yamagata lineage)-like virus strain.
Proportion of participants who do not achieve seroprotection for any influenza virus strains | Week 8
  Seroprotection is defined as HAI titre of ≥1:40
Seroprotection for 1 influenza virus strain | Week 8
  The proportion of participants achieving seroprotection (HAI titre of ≥1:40) for 1 influenza virus strain.
Seroprotection for 2 influenza virus strains | Week 8
  The proportion of participants achieving seroprotection (HAI titre of ≥1:40) for 2 influenza virus strains.
Seroprotection for 3 influenza virus strains | Week 8
  The proportion of participants achieving seroprotection (HAI titre of ≥1:40) for 3 influenza virus strains.
Seroprotection for 4 influenza virus strains | Week 8
  The proportion of participants achieving seroprotection (HAI titre of ≥1:40) for all 4 influenza virus strains.
Markers of immunological function | Week 0, 4 and 8
  Isolation of peripheral blood mononuclear cells (PBMCs) to assess markers of immunological function.
Incidence of upper respiratory symptoms | Week 4, 8, 12 and 16
  Measured using the Wisconsin Upper Respiratory Symptom Survey (WURSS-24).
Faecal gut microbiota (composition, alpha- and beta-diversity) | Week 0, 4 and 8
  Measured by 16S community profiling (Illumina Miseq) of bacterial genomic DNA isolated from stool samples.
Faecal short-chain fatty acids (SCFA) | Week 0, 4 and 8
  Measured by gas liquid chromatography of stool samples.
Faecal water | Week 0, 4 and 8
  Determined from stool samples by oven-drying.
Gut symptoms | Week 0, 4 and 8
  Measured using the Gastrointestinal Symptom Rating Scale (GSRS) (7-day diary; questionnaire).
Stool frequency | Week 0, 4 and 8
  Measured using self-reported number bowel movements daily recorded in a 7-day diary.
Stool consistency | Week 0, 4 and 8
  Measured using the Bristol stool form scale (7-day dairy; questionnaire).
Serum Vitamin E levels | Week 0, 4 and 8
  Measured in blood sample - analysis of serum vitamin E levels by Liquid chromatography-mass spectrometry.
Serum Zinc levels | Week 0, 4 and 8
  Measured in blood sample - analysis of serum zinc levels by automated assay.
Mental health status | Week 0, 4 and 8
  Measured using The Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS). Scores range from 0-48 with higher scores indicating more severe depression/anxiety.
Dietary intake | Week 0, 4 and 8
  7-day food and drink diary.
Physical activity | Week 0, 4 and 8
  Measured using the International Physical Activity Questionnaire (IPAQ).
Acceptability of snack products | Week 8
  Measured using an Acceptability of dietary intervention questionnaire developed by King's College London for use in dietary intervention studies. The questionnaire assesses acceptability using a number of domains including flavour, texture, portion size.
Compliance | Week 8
  Return of unused snacks at the final visit (consumption of >75% of total snacks will be considered compliant).
Adverse events | Week 0 - 8
  Interview-administered questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No